CLINICAL TRIAL: NCT06375356
Title: Stronger: Muscle Strengthening for Menopause
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Marily Ann Oppezzo, Instructor, Med/Stanford Prevention Research Center, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 75119
Record Dates: First submitted 2024-04-12; First posted 2024-04-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Resistance Training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shorter Resistance Training: Stronger Snacks (Experimental): Home-based strength training exercises would be broken up into shorter segments throughout the day or week (e.g. a "snack" might be 3 sets of body-weight or band-based squats).
  Interventions: Behavioral: Resistance Training
- Single Session Resistance Training: Stronger Sessions (Experimental): Home-based strength training exercises would be broken up into 3 weekly sessions throughout the week.
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training — Strength exercises (3-4 sets each exercise) videos delivered electronically, participant self-tracks and self-progresses based on effort reported.

SUMMARY:
Menopause is a period of time with increased risk for muscle and bone loss. Very few people strength train regularly at least 2 times per week, and commonly reported barriers include inadequate time and resources, worries of safety, inadequate knowledge base of what moves to do and how to do them. Menopause-aged women may report unique barriers - or perceived facilitators - to strength training. This pilot study will develop and test the feasibility and acceptability of an at-home, band-based, expert-supported strength training intervention.

DETAILED DESCRIPTION:
Women are at particular risk for low muscle mass as they age, because menopause causes a dramatic reduction in circulating estrogen, which accelerates muscle decline. Preserving muscle is one of the single most important factors to maintaining lifelong independence, with bone, metabolic, cardiovascular, and cognitive health benefits. The most critical behavior for growing and preserving muscle is resistance training, and conservative estimates indicate 4 in 5 US adults do not engage in any resistance training. Commonly cited barriers for women include gender-based stigmas, discouragement, negative comments, poor knowledge of how to do resistance training, poor gym accessibility, and difficulty balancing work and family life. Finally, many menopause practitioners note that with bodyweight as a large concern, many women decrease calorie intake and increase cardiovascular (not resistance) training, further compounding muscle loss. This proposed intervention study aims to develop and pilot a muscle health building intervention with and for menopausal women.

Broadly, the investigators will identify the adherence, feasibility, acceptability, and preliminary changes of a resistance training intervention for menopausal women. The investigators will pilot the 3-month "Stronger" intervention, utilizing a protocol co-designed from focus groups. We will recruit women with menopause and randomize them into one of 2 groups: 1) single-session strength training (Stronger); or 2) "Stronger snacks," the same exercises as the single-session training but broken into single-set snack sizes that are performed throughout the week. The investigators hypothesize that the strength snacks will have the highest adherence and be the most behaviorally accessible and acceptable, but post-study interviews will also help us identify motivational differences.

ELIGIBILITY:
Inclusion Criteria:

* one year of no periods or categorized as menopause
* female at birth
* English speaking

Exclusion Criteria:

* unable to perform strength training movements
* currently performing regular strength training activities or exercise

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
number of strength exercises the participant logged over the intervention | Total at the end of 3 months
  The total number of strength exercises the participant logs is a measure of adherence to the intervention.
Liking of the intervention | 3 month
  Liking is measured using a 5-point Likert scale from not at all (1) to extremely (5) at the end of the intervention as a measure of acceptability of the intervention.

SECONDARY OUTCOMES:
Number of participants completing post 3 month measure / those randomized and consented | 3 months
  This measures retention rate; this will be a single ratio determined by the denominator of number of participants randomized and consented collected at baseline, and a numerator of the number of participants who complete post 3 month measures
Change in total seconds a participant can remain in a wall sit | Change from baseline to 3 months
  This measures muscular strength endurance. Each participant will be timed using a video- when they initiate and when they stop maintaining a position of sitting at 90 degrees with their back supported by the wall behind them.
Change in number of full body weight squats in 60 seconds | Change from baseline to 3 months
  This measures muscular strength endurance. Each participant will video themselves doing bodyweight squats to reach a chair with a bell on it. Each time they touch the bell will count as a rep.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available after publication of primary outcomes of the pilot study.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: After the primary outcomes of this pilot have been published, deidentified data will be available upon request.
Access Criteria: proposed use of the data requested is required